CLINICAL TRIAL: NCT04165629
Title: Influence of Platelet Reactivity in Peripheral Arterial Disease Patients Undergoing Percutaneous Angioplasty on Mid-term Outcomes
Brief Title: Platelet Reactivity in PAD Undergoing Percutaneous Angioplasty
Acronym: PAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Clinical Centre of Serbia (Other)
Responsible Party: Principal Investigator, Petar Zlatanovic, Medical Doctor, Clinical Centre of Serbia
Other Study IDs: Platelet reactivity in PAD
Record Dates: First submitted 2019-11-14; First posted 2019-11-18 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Peripheral Artery Disease; Critical Limb Ischemia; Claudication, Intermittent
MeSH Terms: conditions — Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia; Intermittent Claudication | interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Aspirin responders: On impedance aggregometry- Multiplate analyzer, if ASPI < 600 or ASPI/TRAP < 0.5
  Interventions: Drug: Aspirin 300mg and Clopidogrel 300mg
- Aspirin non-responders: On impedance aggregometry- Multiplate analyzer, if ASPI > 600 or ASPI/TRAP > 0.5
  Interventions: Drug: Aspirin 300mg and Clopidogrel 300mg
- Clopidogrel responders: On impedance aggregometry- Multiplate analyzer, if ADP < 500 or ADP/TRAP < 0.5
  Interventions: Drug: Aspirin 300mg and Clopidogrel 300mg
- Clopidogrel non-responders: On impedance aggregometry- Multiplate analyzer, if ADP > 500 or ADP/TRAP > 0.5
  Interventions: Drug: Aspirin 300mg and Clopidogrel 300mg

INTERVENTIONS:
Drug: Aspirin 300mg and Clopidogrel 300mg — Aspirin 300mg and Clopidogrel 300mg on the day of the PTA

SUMMARY:
Dual antiplatelet therapy has a key role in a prevention of thrombosis of treated artery in patients undergoing percutaneous transluminal angioplasty (PTA). Weak therapeutic response and presence of residual platelet activity is related to high risk for stent thrombosis and it is well in known in coronary artery disease (CAD) patients undergoing percutaneous coronary intervention (PCI). However there are few data on the association between a different entity of platelet inhibition on antiplatelet treatment and clinical outcomes in patients with peripheral artery disease (PAD). The aim of this study was to evaluate the degree of on-treatment platelet reactivity, and its association with ischemic and hemorrhagic adverse events at follow up in PAD patients undergoing PTA.

DETAILED DESCRIPTION:
This is a single-center observational cohort study. All together 450 patients undergoing and elective PTA (both with and without stenting) who are going to be refereed to the Clinic for Vascular and Endovascular Surgery (based on the previous experience) during the two year period (January 1st 2020 and January 1st 2022) are planned to be involved in this study. All interventions will be performed according to the current standards and the type of the endovascular procedure will be at the discretion of operator. All patients will receive at the day of treatment 300mg of Aspirin and 300mg of Clopidogrel. The day after the procedure platelet function will be assessed by "point-of-care" impedance aggregometry test using the Multiplate analyzer. According to the manufacturer proposition, resistancy on Aspirin will be defined as arachidonic acid receptor (ASPI) value < 600 and ASPI/thrombin receptor activating peptide (TRAP) < 0.5, and for Clopidogrel adenosine diphosphate (ADP) < 500 and ADP/TRAP < 0.5 . After that patients will receive dual antiplatelet therapy (Aspirin 100mg and Clopidogrel 75mg) in the six months period. Follow-up examinations will be scheduled on 1, 6 and 12 months after the intervention. Adherence to antiplatelet treatment will assessed during scheduled or unscheduled examinations. Statistical analysis will be performed using the software package SPSS 20 (SPSS Inc., Chicago, Il, USA). Categorical data will be represented as numbers and percentages. Chi-square test or Fisher exact test as appropriate will be used to compare categorical data. Continuous variables will be represented as mean ± standard deviation and as median and interquartile range, depending on the normality of data. Student's t test or Mann-Whitney U test as appropriate will be used to compare two population groups. We will then assess the ability of ASPI and ADP values to distinguish between patients with and without clinical event at 6 months follow up by receiver-operating characteristic (ROC) curve analysis and the optimal cut-off ASPI and ADP values will be determined by estimating the value resulting in the maximum sum of sensitivity and specificity (area under the curve - AUC). Kaplan-Meier curves with log-rank test will be used to assess difference in the time-to-event end-points. A multivariable Cox proportional hazard model adjusted for clinical and laboratory variables will be performed to evaluate the independent contribution of platelet hyper- or hypo-reactivity to the outcomes. A P-values <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

- all patients treated due to PAD with PTA with/without stenting of aorto-iliac, femoro-popliteal and crural disease at the mentioned time period with critical limb ischemia (CLI) or intermittent claudication (IC)

Exclusion Criteria:

* younger that 18 and older than 85
* contraindications for Aspirin and Clopidogrel use
* thrombocytopenia (<100 x 10⁹/l)
* thrombocytosis (>450 x 10⁹/l)
* kidney insufficiency (stage 4 and 5)
* more severe anemia (Hgb < 100 g/l)
* severe hepatic disorder
* congestive heart failure
* known hemorrhagic disorder
* known malignant disease
* previous use of drugs with known anti-thrombocyte mechanism of action (dipyridamole, NSAID)
* use oral anticoagulant therapy
* use of corticosteroids
* use of drugs that are metabolized threw CYP3A4 (like erythromycin and rifampicin)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated at the Clinic for Vascular and Endovascular Surgery, Clinical Center of Serbia, Belgrade due to PAD (critical limb ischemia {CLI} or intermittent claudication {IC}) with PTA with/without stenting of aorto-iliac, femoro-popliteal and crural disease between January 1st 2020 and January 1st 2022
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Limb Event (MALE) | 6 months
  It includes major amputation, reintervention which could be surgical or repeat angioplasty. Major amputation is defined as amputation above the ankle.
Mortality | 6 months
  All-cause mortality

SECONDARY OUTCOMES:
Major Adverse Cardio- and Cerebrovascular Events (MACCE) | 6 months
  Nonfatal stroke, nonfatal myocardial infarction, and cardiovascular death
Bleeding complications | 6 months
  Major and minor bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Petar Zlatanovic, MD, Principal Investigator — Clinical Center of Serbia
Locations (1):
- Clinical Center of Serbia, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: Undecided
to be available on request for now

REFERENCES:
- [Background] Spiliopoulos S, Pastromas G, Katsanos K, Kitrou P, Karnabatidis D, Siablis D. Platelet responsiveness to clopidogrel treatment after peripheral endovascular procedures: the PRECLOP study: clinical impact and optimal cutoff value of on-treatment high platelet reactivity. J Am Coll Cardiol. 2013 Jun 18;61(24):2428-2434. doi: 10.1016/j.jacc.2013.03.036. Epub 2013 Apr 16. PMID 23602777
- [Background] Grifoni E, Gori AM, Giusti B, Valenti R, Migliorini A, Basili S, Paniccia R, Elmahdy MF, Pulli R, Pratesi C, Antoniucci D, Violi F, Marcucci R. On-Treatment Platelet Reactivity is a Predictor of Adverse Events in Peripheral Artery Disease Patients Undergoing Percutaneous Angioplasty. Eur J Vasc Endovasc Surg. 2018 Oct;56(4):545-552. doi: 10.1016/j.ejvs.2018.06.032. Epub 2018 Jul 17. PMID 30025662
- [Background] Leunissen TC, Peeters Weem SM, Urbanus RT, den Ruijter HM, Moll FL, Asselbergs FW, de Borst GJ. High On-Treatment Platelet Reactivity in Peripheral Arterial Disease: A Pilot Study to Find the Optimal Test and Cut Off Values. Eur J Vasc Endovasc Surg. 2016 Aug;52(2):198-204. doi: 10.1016/j.ejvs.2016.04.019. Epub 2016 May 25. PMID 27236738
- [Background] Pastromas G, Spiliopoulos S, Katsanos K, Diamantopoulos A, Kitrou P, Karnabatidis D, Siablis D. Clopidogrel responsiveness in patients undergoing peripheral angioplasty. Cardiovasc Intervent Radiol. 2013 Dec;36(6):1493-1499. doi: 10.1007/s00270-013-0577-3. Epub 2013 Feb 14. PMID 23408060
- [Background] Spiliopoulos S, Pastromas G. Current status of high on-treatment platelet reactivity in patients with coronary or peripheral arterial disease: Mechanisms, evaluation and clinical implications. World J Cardiol. 2015 Dec 26;7(12):912-21. doi: 10.4330/wjc.v7.i12.912. PMID 26730297